CLINICAL TRIAL: NCT07248514
Title: Effects of Pilates on Pain and Trunk Muscle Endurance in Children With Backpack Syndrome
Brief Title: Effect of Pillates on Children With Backpack Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/MUHAMMADFAROOQI
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Child, Only
Keywords: Pilates, Modified Biering-Sørensen Test
MeSH Terms: interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: This randomized clinical trial focuses on a sample of 140 of children diagnosed with backpack syndrome, assessing both subjective pain levels and objective measures of trunk muscle endurance before and after a structured Pilates intervention. The Pilates regimen is designed to strengthen core muscles, improve flexibility, and promote better posture, all of which are critical for mitigating the adverse effects associated with heavy backpack use.Data will be collected from North Star School Allama Iqbal town,Lahore,Standard Grammar School, Allama iqbal town ,Kips School, Allama iqbal town,Ali School System, Allama Iqbal Town Using standardized pain assessment scales(VAS) and endurance tests(Modified Biering-Sørensen Test), the effect of pilates on pain and trunk endurance will concluded and the data will analysed with spss 23.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Interventional group
  Interventions: Other: Pilates exercise
- Group B (Active Comparator): Experimental group
  Interventions: Other: General Stretching exercises

INTERVENTIONS:
Other: Pilates exercise — The exercise program will be performed twice a week for 12 weeks changing the exercises for every four weeks. Pilates exercises will consist of four exercises which are selected from original Pilates plan (month 1: rolling back, one leg stretch, shoulder bridge and the push up; month 2: the hundred, one leg stretch, the leg pull and one leg circle; month 3: roll up, scissors, swimming and one leg stretch) (4)
  Arms: Group A
Other: General Stretching exercises — Group B will perform routine physical therapy (RPT) alone. These routine exercises will consist of stretching exercises adding some games, stretching and relaxation exercises at the end. i,e stretching exercises, posture training, and spinal flexibility exercises
  Arms: Group B

SUMMARY:
This randomized clinical trial focuses on a sample of 139 of children diagnosed with backpack syndrome, assessing both subjective pain levels and objective measures of trunk muscle endurance before and after a structured Pilates intervention. The Pilates regimen is designed to strengthen core muscles, improve flexibility, and promote better posture, all of which are critical for mitigating the adverse effects associated with heavy backpack use.Data will be collected from North Star School Allama Iqbal town,Lahore,Standard Grammar School, Allama iqbal town ,Kips School, Allama iqbal town,Ali School System, Allama Iqbal Town Using standardized pain assessment scales(VAS) and endurance tests(Modified Biering-Sørensen Test), the effect of pilates on pain and trunk endurance will concluded and the data will analysed with spss 23

DETAILED DESCRIPTION:
The research titled "Effects of Pilates on Pain and Trunk Muscle Endurance in Children with Backpack Syndrome" investigates the impact of Pilates exercises on alleviating pain and enhancing trunk muscle endurance in children affected by backpack syndrome. Backpack syndrome refers to musculoskeletal discomfort resulting from improper backpack use, often seen in school-aged children who carry heavy loads, leading to poor posture and potential long-term health issues.

This randomized clinical trial focuses on a sample of 139 of children diagnosed with backpack syndrome, assessing both subjective pain levels and objective measures of trunk muscle endurance before and after a structured Pilates intervention. The Pilates regimen is designed to strengthen core muscles, improve flexibility, and promote better posture, all of which are critical for mitigating the adverse effects associated with heavy backpack use.Data will be collected from North Star School Allama Iqbal town,Lahore,Standard Grammar School, Allama iqbal town ,Kips School, Allama iqbal town,Ali School System, Allama Iqbal Town Using standardized pain assessment scales(VAS) and endurance tests(Modified Biering-Sørensen Test), the effect of pilates on pain and trunk endurance will concluded and the data will analysed with spss 23.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 12-16 years.
* Being Systemically healthy
* Being physically active and participating in ordinary assessments(4)
* Children with musculoskeletal backpain
* Children with hyper thoracic kyphosis i.e. excessive antero-posterior curvature of the thoracic spine of greater than 40°
* Children complaining about low back pain

Exclusion Criteria:

* Children with a history of severe musculoskeletal conditions (e.g., scoliosis, fractures, or surgery).
* Any neurological disorders or developmental conditions affecting motor function
* Children with cardiological, metabolic or rheumatic illness
* Children with no complaints of low back pain and postural instability.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analouge Scale | 12 weeks
  The Visual Analog Scale (VAS) is a tool used to measure subjective characteristics or attitudes that cannot be directly measured, commonly used in pain assessment. The scale is often represented as a horizontal line, typically 10 cm in length, anchored by terms at each end that represent extremes of the sensation being measured
Modified Biering-Sørensen | 12 weeks
  The Modified Biering-Sørensen Test is an adaptation of the original Biering-Sørensen test, used to assess endurance in the muscles of the lower back, particularly the lumbar extensor muscles. The test measures how long a person can hold a specific static position, which helps evaluate core strength and endurance.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Farooqi, MS-PT, Principal Investigator — Riphah International University
Locations (1):
- Imran Amjad, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gonzalez-Galvez N, Vaquero-Cristobal R, Marcos-Pardo PJ. Effect of Pilates Method on muscular trunk endurance and hamstring extensibility in adolescents during twelve weeks training and detraining. J Bodyw Mov Ther. 2020 Apr;24(2):11-17. doi: 10.1016/j.jbmt.2020.02.002. Epub 2020 Feb 21. PMID 32507135